CLINICAL TRIAL: NCT02597179
Title: Genome Sequencing in Refractory Breast Cancer to Molecular Targeted Therapy and Young Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, MD, Ph.D, Division of Hematology-Oncology, Samsung Medical Center
Other Study IDs: 2012-08-065
Record Dates: First submitted 2015-10-29; First posted 2015-11-05 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Breast Cancer, Young Breast Cancer: Patients with feasible biopsy site.

SUMMARY:
The purpose of this study is to investigate and analyse genomic profiles in patient with breast cancer who failed standard treatment, refractory and young breast cancer.

DETAILED DESCRIPTION:
The hypothesis is that genomic profiling measured by CancerSCAN, cfDNA, Whole exome sequencing (WES), Whole transcriptome sequencing (WTS), FACS(Fluorescence-Activated Cell Sorting), cytokine and immunologic signature analysis would be helpful to find out tolerance for chemotherapy and innovate new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed breast cancer that is either metastatic or young breast cancer(≤ 40 years of age).
2. HER2 positive patient who failed HER2 target therapy including trastuzumab with feasible biopsy site.
3. Triple Negative Breast Cancer patient who failed standard therapy with feasible biopsy site.
4. Hormone Receptor positive patient who failed standard therapy with feasible biopsy site.
5. Age ≥ 21 years
6. Written informed consent

Exclusion Criteria:

1. No feasible biopsy site
2. No written informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically conrfirmed breast cancer that is either metastatic or young breast cancer(≤ 40 years of age) with feasible biopsy site.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Mutated Genes and/or Abnormal Gene expression and/or Different Immune signature That Affect to Treatment Outcome. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-Gu, South Korea